CLINICAL TRIAL: NCT02317965
Title: A Prospective Clinical Study to Evaluate a Novel Non-invasive Prenatal Screening Method for Characterizing Fetal Whole Chromosome Aberrations and Other Major Defects and Deletions Found in the Maternal Blood.
Brief Title: Non-Invasive Screening for Fetal Aneuploidy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Progenity, Inc. (Industry)
Collaborators: Obstetrix Medical Group (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-100
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Down Syndrome; Edwards Syndrome
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Pregnant women who are scheduled to undergo an amniocentesis or chorionic villus sampling (CVS) procedure
  Intervention: Single Maternal blood draw of 20mL
  Interventions: Other: Maternal Blood Draw

INTERVENTIONS:
Other: Maternal Blood Draw — Maternal Blood Draw

SUMMARY:
The purpose of this study is to detect whole chromosome abnormalities in maternal blood.

DETAILED DESCRIPTION:
The purpose of this study is to detect whole chromosome abnormalities on all chromosomes 13, 16, 18, 21, X and Y, in the fetus through analysis of cell free and compound sample DNA (cf DNA and cs DNA, respectively) in maternal blood. In addition, major deletions and duplications in chromosomes 1, 4, 5, and 22 will be detected.

ELIGIBILITY:
Inclusion Criteria:

* • Subject is a pregnant woman 18-54 years of age at 8-22 weeks' gestation inclusive;

  * Subject has additional risk indicators for fetal chromosome aneuploidy, including one or more of the following:
  * Maternal age > 34 years at the estimated date of delivery;
  * Positive serum screening test suggesting fetal aneuploidy;
  * Previous positive noninvasive cfDNA test is acceptable
  * Fetal ultrasound abnormality suggesting fetal chromosomal abnormality;
  * Personal or family history of Down syndrome or other chromosomal aneuploidy.
  * Willing to provide written informed consent
  * Willing to be re-contacted subsequently for additional information and/or testing if necessary.

Exclusion Criteria:

* Subjects will not be entered into this study if they meet the following criteria:

  * Fetal demise at the time of the blood draw;
  * Previous specimen donation under this protocol;
  * Unwilling or lacks the capacity to provide informed consent or to comply with study procedures;
  * Currently under treatment for cancer
  * Any history of autoimmune disease
  * Any pelvic mass
  * Previous history of radiation to pelvis
  * Any history or current evidence of a twin demise at any gestational age.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women who are scheduled to undergo an amniocentesis or CVS procedure and will receive the fetal FISH and/or karyotype results from the procedure.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Validate the prenatal aneuploidy laboratory developed test (LDT) with maternal blood samples from pregnant women who are undergoing invasive prenatal diagnosis | Participants will have a single visit and completion in study occurs once invasive procedure results have been recorded.
  A single 20 mL blood sample will be obtained from each subject during the first or second trimester, blind-coded, and transferred to the Sponsor Laboratory for processing to plasma.
  Subjects electing to undergo an invasive procedure for fetal Karyotyping (defined as standard cytogenetics and/or microarray, FISH, QF-PCR) will have the blood sample obtained prior to the procedure.
  The performance characteristics (sensitivity, specificity, negative and positive predictive value) of the laboratory developed test to detect whole chromosome abnormalities on all chromosomes 13, 16, 18, 21, X and Y will be determined using fetal karyotype on specimens obtained by chorionic villus sampling and/or genetic amniocentesis for those subjects who undergo these diagnostic procedures as part of their standard care as the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Porreco, MD, Principal Investigator — Obstetrix Medical Group of Colorado; Thomas Garite, MD, Study Director — Obstetrix Medical Group
Locations (10):
- United States (10):
  - Obstetrix Medical Group of California, Campbell, California
  - Long Beach Memorial Medical Ctr - 2nd Floor Perinatal, Long Beach, California
  - OBX Med. Group. of Colorado - Pres/St Luke's Clinic, Denver, Colorado
  - OBX Med. Group. of Colorado - Antepartum Testing Unit @ Rose Medical Center, Denver, Colorado
  - OBX Med. Group. of Colorado - Perinatal Resource Ctr @ Swedish Med Ctr., Englewood, Colorado
  - OBX Med. Group. of Colorado - Skyridge, Lone Tree, Colorado
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - Obstetrix Medical Group of Texas, Fort Worth, Texas
  - Obstetrix Medical Group of Houston, The Woodlands, Texas
  - Obstetrix, Medical Group of Washington, Inc. - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Porreco RP, Sekedat M, Bombard A, Garite TJ, Maurel K, Marusiak B, Adair D, Bleich A, Combs CA, Kramer W, Longo S, Nageotte M, Samuel A, Vanderhoeven J, Buis J, Jacobs KB, Stoerker J. Evaluation of a novel screening method for fetal aneuploidy using cell-free DNA in maternal plasma. J Med Screen. 2020 Mar;27(1):1-8. doi: 10.1177/0969141319873682. Epub 2019 Sep 11. PMID 31510865